CLINICAL TRIAL: NCT06076135
Title: Efficacy and Safety of Combining Intestinal Low Dose Radiotherapy and PD-1/PD-L1 Inhibitors for Metastatic Malignant Solid Tumors After Acquired Resistance to Anti-PD1/PD-L1 Treatment
Brief Title: Intestinal Low Dose Radiotherapy Combined With Immunotherapy in Immune-resistant Metastatic Solid Tumors
Acronym: ILDR-01
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chuangzhen Chen (Other)
Responsible Party: Sponsor-Investigator, Chuangzhen Chen, Dr, Shantou University Medical College
Organization: Shantou University Medical College (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ShantouUMC
Record Dates: First submitted 2023-09-28; First posted 2023-10-10 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Metastatic Malignant Solid Neoplasm; Radiotherapy; Immune Checkpoint Blockade; Resistance to Immunotherapy
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Stage Ⅰ (Experimental): 1Gy/1F ILDR + PD-1/PD-L1 inhibitors.
  Interventions: Radiation: Intestinal Low Dose Radiotherapy-1Gy; Drug: PD-1/PD-L1 Inhibitors
- Treatment Stage Ⅱ (Experimental): 2-3Gy/2-3F ILDR + PD-1/PD-L1 inhibitors.
  Interventions: Radiation: Intestinal Low Dose Radiotherapy-2-3Gy; Drug: PD-1/PD-L1 Inhibitors

INTERVENTIONS:
Radiation: Intestinal Low Dose Radiotherapy-1Gy — 1Gy ILDR will be administered to patients in a single fraction. The radiation treatment volume composes both the jejunum and ileum.
  Arms: Treatment Stage Ⅰ
Radiation: Intestinal Low Dose Radiotherapy-2-3Gy — ILDR will be administered as single fractions within 10 days. The total dose of radiotherapy will be 2-3 Gy in 2-3 fractions. ILDR design is as above.
  Arms: Treatment Stage Ⅱ
Drug: PD-1/PD-L1 Inhibitors — The immunotherapy regimen is the previous ICB therapy regimen or modified by the physician in charge. PD-1/PD-L1 inhibitors will be given 1 day after ILDR at a 3-week interval.

SUMMARY:
Preclinical and clinical studies have shown that intestinal low dose radiotherapy (ILDR) can enhance antitumor immunity and response to immune checkpoint blockade (ICB). Therefore, the investigators launch a phase Ⅱ trial to evaluate the clinical value of combining ILDR and programmed cell death-1/ -ligand 1 (PD-1/PD-L1) inhibitors in patients with ICB refractory metastatic solid tumor.

This study is designed as a researcher-initiated, two-stage and prospective clinical trial. The target population is patients with advanced metastatic malignant solid tumors who have progressed after immunotherapy. The primary endpoints include objective response rate (ORR), disease control rate (DCR), progression free survival while receiving ILDR combined therapy (PFS2), and lesion-based abscopal response rate. The secondary endpoints include incidence of adverse events (AEs), cancer-specific survival (CSS), and overall response rate (OS).

In the treatment stage Ⅰ, sixteen subjects will be enrolled in this trial. The primary objective of this stage is to evaluate the safety and efficacy of 1Gy ILDR combined with PD-1/PD-L1 inhibitors in immune-resistant metastatic malignant solid tumors, and biomarker exploration for response prediction.

The inclusion criteria, exclusion criteria and sample size for treatment stage Ⅱ will be modified on the basis of results from Stage Ⅰ. The objective of the stage Ⅱ is to determine effects and safety of various dosage regimen of ILDR combined with PD-1/PD-L1 inhibitors in target patients.

Eligible patients will be subjected to 1-3Gy ILDR. Tumor response will be assessed according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 as well as Immune related RECIST (iRECSIST). The extent or severity of adverse reactions will be assessed using Common Terminology Criteria for Adverse Events (CTCAE) (version 5.0). Furthermore, tissue samples, stool samples, and peripheral blood samples will be collected for biomarker exploration.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, ≤80 years, regardless of gender.
2. ECOG level 0-2.
3. Expected life span>3 months.
4. At least one accessible and measurable lesion should be selected as the target lesion for observation according to RECIST criteria.
5. Patients with metastatic solid tumors (of any histology) without standard therapy options, who have previously received immunotherapy, immunotherapy combined with chemotherapy, or immunotherapy combined with anti-angiogenesis treatment and have shown disease progression.
6. The patient is considered ineligible for surgical treatment.
7. Patients with brain metastases assessed as clinically stable after treatment through repeated CT and/or MRI scans are eligible.
8. Patients have complete clinical and pathological information.
9. Any psychological, family, social or geographical conditions may hinder compliance with the research protocol.
10. Patients are able to understand the informed consent form, voluntarily participate, and sign the informed consent form.
11. Other indicators accord with the general inclusion criteria for clinical trials.

Exclusion Criteria:

1. Patients with contraindications to radiation therapy and immunotherapy.
2. Previous occurrence of unacceptable immune related toxic side effects (immune myocarditis, pneumonia, etc.).
3. Patients who were assessed as hyperprogressive disease (HPD).
4. Patients who have received pelvic and abdominal radiation therapy within 6 months prior to enrollment.
5. The adverse reactions from prior treatment have not yet recovered to a CTCAE5.0 rating of ≤ 1 (excluding toxicity that has been determined to be risk-free, such as fatigue or hair loss).
6. Accompanied by severe infections.
7. Serious liver disease (such as cirrhosis), kidney disease, respiratory disease, or chronic system diseases such as uncontrollable diabetes and hypertension; Patients who cannot tolerate radiation therapy.
8. Clinical symptoms of brain metastases or meningeal metastasis.
9. The patients with known allergies or allergies to the test drug ingredients.
10. Substance/alcohol abuse.
11. Patients who are pregnant or planning to.
12. Patients participating in other clinical studies that may affect the efficacy/safety of this clinical study.
13. Patients who have undergone major surgical procedures within 30 days.
14. Patients who have received antibiotics, antifungal drugs, antiviral, antiparasitic drugs, or probiotics within 4 weeks.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-12-26 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 6, 12, 24 weeks after start of ILDR.
  The objective effective rate of ILDR combined with PD-1/PD-L1 inhibitors in patients with metastatic malignant solid tumors after acquired resistance to immunotherapy, including complete response and partial response.
Disease Control Rate（DCR） | 6, 12, 24 weeks after start of ILDR.
  The proportion of patients with optimal response to ILDR combined with PD-1/PD-L1 inhibitors.
Progression Free Survival while Receiving ILDR combined Therapy (PFS2) | 6, 12, 24 weeks after start of ILDR.
  The time from the date of ILDR initiation to the documented disease progression or death due to cancer.
Lesion-based Abscopal Response Rate | 6, 12, 24 weeks after start of ILDR.
  The proportion of patients with tumor objective response in one or more lesions.

SECONDARY OUTCOMES:
Incidence of Adverse Events | 12, 24, 48 weeks after start of ILDR.
  The proportion of patients with treatment-related adverse events as assessed by CTCAE v5.0.
Overall survival (OS) | 24, 48 weeks after start of ILDR.
  The time from the date of ILDR initiation to death from any cause.
Cancer-specific survival (CSS) | 24, 48 weeks after start of ILDR.
  The time from the date of ILDR initiation to death due to cancer.

OTHER OUTCOMES:
Changes of Intestinal Flora | Before the first treatment, 3-7 days after start of ILDR, before each immunotherapy.
  Fecal samples are analyzed by metagenomics sequencing. The differential intestinal flora is obtained through differential analysis, and the correlation between the differential microbial communities and other indicators is analyzed.
Metabolites in fecal samples | Before the first treatment, 3-7 days after start of ILDR, before each immunotherapy.
  The wide arrays of metabolites in fecal samples are analyzed qualitatively and quantitatively.
Tissue Immune Analyses | Before the first treatment, 3 weeks after start of ILDR.
  Tumor tissue is obtained for histopathological staining and transcriptome sequencing.
Peripheral Blood Immune Analyses | Before the first treatment, 3-7 days after start of ILDR, before each immunotherapy.
  Flow cytometry analysis is performed on peripheral blood samples.
Changes of Serum Metabolites | Before the first treatment, 3-7 days after start of ILDR, before each immunotherapy.
  The wide arrays of metabolites in serum are analyzed qualitatively and quantitatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital, Shantou University Medical College, Shantou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No